CLINICAL TRIAL: NCT01167803
Title: Coming Out of Anesthesia After Bariatric Surgery : Desflurane Versus Xenon
Brief Title: Anesthesia for Obese Patients: Desflurane Versus Xenon
Acronym: XENON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC-I/2009/EN-01; 2009-017126-39 (EudraCT Number)
Record Dates: First submitted 2010-07-21; First posted 2010-07-22 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
Keywords: Bariatric surgery; Anesthesia
MeSH Terms: conditions — Obesity | interventions — Desflurane; Xenon

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Reference - desflurane (Active Comparator): The patients in this group will undergo anesthesia using remifentanil associated with desflurane.
  Interventions: Drug: Desflurane
- Experimental - xenon (Experimental): The patients in this group will undergo anesthesia using remifentanil associated with xenon
  Interventions: Drug: Xenon

INTERVENTIONS:
Drug: Desflurane — Patients undergo anesthesia using remifentanil associated with desflurane
  Arms: Reference - desflurane
Drug: Xenon — Patients undergo anesthesia using remifentanil associated with xenon
  Arms: Experimental - xenon

SUMMARY:
Obesity is increasing in France, resulting in an increased demand for bariatric surgery. However obesity also alters physiopathological pathways and the pharmacokinetics of anesthestic agents. The investigators objective is to compare, among morbidly obese patients, the immediate and intermediary emergence kinetics after balanced anesthesia using remifentanil associated either with desflurane (reference arm) or with xenon (experimental arm).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) I to III
* requires bariatric surgery
* body mass index (BMI) >= 35 kg/m2
* patient speaks and writes French
* patient has signed consent form
* patient enrolled in a social security program

Exclusion Criteria:

* patient refuses to sign consent
* ASA IV or more
* patient is pregnant or breastfeeding
* history of hyperthermy (or suspicion, or family history thereof)
* history of liver disease, icterus, unexplained fever, or eosinophilia after administration of a halogen anesthesia
* patient has symptomatic gastro-oesophagean reflux
* patient has hypersensitivity to one or more of the following substances: propofol, remifentanil, celocurine, cisatracurium, rocuronium, desflurane, xenon, paracetamol, ketoprofen, nefopam, tramadol
* patient has obstructive respiratory failure (chronic obstruction pneumopathy, asthma) or has heart disease with severly altered cardiac function
* patient has high intracranial pressure
* patient requires high concentrations of oxygen (fio2>40%)
* patient has a neuro-sensorial deficient which prevents reading, writing, or response to simple oral commands (severe deafness, language impairment...)in the absence of a prothesis
* patient has a psychiatric pathology, or chronically consumes alcohol or other mind-altering substance
* patient has had general anesthesia in the last 15 days
* patient under guardianship
* impossible to correctly communicate information to the patient
* absence of efficient contraception for women of childbearing age
* participation in another study within the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2010-12; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
30 min DSST ratio | 30 minutes post-op
  (the number of correct responses to a Digit Symbol Substitution Test [DSST] 30 minutes after surgery) / (the number of correct responses to a Digit Symbol Substitution Test the night before the surgery)

SECONDARY OUTCOMES:
60 min DSST test | 60 minutes post-op
  (the number of correct responses to a Digit Symbol Substitution Test 60 minutes after surgery) / (the number of correct responses to a Digit Symbol Substitution Test the night before the surgery)
90 min DSST test | 90 min post-op
  (the number of correct responses to a Digit Symbol Substitution Test 90 minutes after surgery) / (the number of correct responses to a Digit Symbol Substitution Test the night before the surgery)
Time to Aldrete score of 10 | Immediate post-op; this outcome measures the minutes of emergence (from anesthesia) time necessary to attain an Aldrete score of 10
  Aldrete JA. The post-anesthesia recovery score revisited. J. Clin. Anesth. 1995.
Quality of recovery score | Day 1 post-op
  The score on the Quality of Recovery Scale:
  Myles PS, Weitkamp B, Jones K et al. Validity and reliability of a postoperative quality of recovery score: the QoR-40. Br. J. Anaesth., 2000; 84: 11-15.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Ripart, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (6):
- France (6):
  - CHU de Clermont Ferrand - Hôpital Estaing, Clermont-Ferrand
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHU de Montpellier - Hôpital Saint-Eloi, Montpellier
  - CHU de Nice - Hôpitaux L'Archet 1 et 2, Nice
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CHU de Poitiers, Poitiers